CLINICAL TRIAL: NCT05604027
Title: The Effects of Pain Types on Pain Severity and Quality of Life in Chronic Low Back Pain
Brief Title: Pain Types and Pain Severity in Chronic Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-15/20
Record Dates: First submitted 2022-10-10; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Visual Analogue Scale — Clinical criteria and rating system for nociplastic pain affecting the musculoskeletal system and PainDETECT scale to determine pain type SF-36 Quality of Life Scale, Roland Morris Disability Questionnaire, Pain Catastrophizing Scale, and Visual Analog Scale to determine the effects
  Other Names: Pain Catastrophizing Scale; The Roland-Morris Disability Questionnaire; Short form-36; painDETECT; Clinical criteria and rating score for nociplastic pain affecting the musculoskeletal system

SUMMARY:
The aim of this study is to characterize the distribution of pain phenotypes in people with chronic low back pain and to determine the effects of pain phenotypes on pain severity, functional status and quality of life.

Participants will be examined to determine the type of pain and questions will be asked to identify the effects.

ELIGIBILITY:
Inclusion Criteria:

* having chronic low back pain
* be over 18 years old

Exclusion Criteria:

* Those under the age of 18
* Those with major psychiatric illness,
* Those with communication problems

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who come to the hospital for chronic low back pain
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
identification of pain types(determination of nociceptive, neuropathic, nociplastic pain rates) | 01.03.2023
  Neuropathic pain with PainDETECT scale, Clinical criteria and rating system for nociplastic pain affecting the musculoskeletal system nosplastic pain will be evaluated
Pain levels of those with nociplastic, neuropathic and nociceptive pain | 01.03.2023
  Pain severity with Visual Analogue Scale,(0-10)higher scores indicate more pain
pain effect | 01.03.2023
  quality of life with SF-36,
disability, | 01.03.2023
  disability with Roland Morris Disability Questionnaire,
patient's feelings, thoughts, and feelings about pain and disaster. | 01.03.2023
  The Pain Catastrophizing Scale is used to assess the patient's feelings, thoughts, and feelings about pain and disaster.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Research and Training Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
will be shared upon request.